CLINICAL TRIAL: NCT02628587
Title: Comparison of Platelet Reactivity in Patients With Acute Coronary Syndrome Given Patent Clopidogrel Versus Generic Clopidogrel: Randomized Controlled Trial
Brief Title: Patent Versus Generic Clopidogrel in Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Central San Luis Potosi, Mexico (Other)
Responsible Party: Principal Investigator, Juan Manuel López Quijano, Dr. Juan Manuel Lopez Quijano, Hospital Central San Luis Potosi, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUZ001
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Clopidogrel; Platelet reactivity
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic clopidogrel (Experimental): Patients are assigned to take generic clopidogrel
  Interventions: Drug: Generic clopidogrel
- Patent clopidogrel (Active Comparator): Patients are assigned to take patent clopidogrel (Plavix)
  Interventions: Drug: Patent clopidogrel

INTERVENTIONS:
Drug: Generic clopidogrel — Comparison of different brands of clopidogrel:
  *Clopidogrel (generic) 300mg orally single dose on day 0. Later, clopidogrel 75mg orally single dose on days 1, 2 and 3.
  Arms: Generic clopidogrel
Drug: Patent clopidogrel — Comparison of different brands of clopidogrel:
  *Clopidogrel (Plavix) 300mg orally single dose on day 0. Later, clopidogrel 75mg orally single dose on days 1, 2 and 3.
  Other Names: Plavix
  Arms: Patent clopidogrel

SUMMARY:
Ischemic heart disease is the leading cause of death and disability in developed countries and is responsible for a third of deaths in persons over 35 years . The most severe form of ischemic heart disease is sudden death and acute coronary syndrome (ACS).

There is evidence that early and optimal treatment of ACS decreases mortality. Within the optimal treatment, these patients must receive a reperfusion therapy as mechanical or pharmacologic treatment. In addition to reperfusion treatment, antiplatelet therapy is a central part of the management. Aspirin plus a P2Y12 inhibitor have been shown to decrease mortality. In our country, clopidogrel is the more accessible and used P2Y12 inhibitor; however, it has been shown to have a wide variability in response and this variability could be influenced by different pharmacological, genetic and environmental factors.

Platelet reactivity measured by aggregometry predicts major cardiovascular events in ACS patients treated with clopidogrel. Due to their frequent prescription, generic clopidogrel efficacy must be evaluated. The purpose of this study is to compare the platelet reactivity in patients with ACS receiving clopidogrel generic versus patent.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Diagnosis of acute coronary syndrome
* Patients receiving 300 mg of Clopidogrel load and a single dose of 75 mg daily
* Signature of informed consent

Exclusion Criteria:

* Active bleeding or absolute contraindication for antiplatelet use
* Chronic kidney disease with creatinine clearance <30 ml / min
* Liver damage documented as elevated aspartate aminotransferase/alanine aspartate 2 times upper normal limit (UNL) and/or total bilirubin > 2 times UNL
* Prescribed antiplatelet therapy, other than aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity change | Day 0 and Day 3
  Change in platelet reactivity measured from day 0 to day 3 of Clopidogrel therapy

IPD SHARING:
Plan to Share IPD: Undecided